CLINICAL TRIAL: NCT04384315
Title: Pilot Study to Investigate the Efficacy and Safety of Endovenous Radio Frequency (EVRF) for Treatment of Varicose Veins in Singapore
Brief Title: Efficacy and Safety of Endovenous Radio Frequency (EVRF) for Treatment of Varicose Veins in Singapore
Acronym: ESVS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2019/2544
Record Dates: First submitted 2020-04-06; First posted 2020-05-12 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Varicose Veins; Venous Reflux; Chronic Venous Insufficiency
Keywords: Endovenous Ablation
MeSH Terms: conditions — Varicose Veins | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EVRF: Patients that have undergone Endovenous Radio Frequency® (EVRF®) from F Care Systems (Belgian) for the treatment of primary great and short saphenous vein reflux.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Questionnaires to assess the quality of life (EQ-5D, CVVQ, CIVIQ, AVVQ, Patient satisfaction survey)

SUMMARY:
The aim of this study is to report a collaborative, prospective Singaporean experience using the Endovenous Radio Frequency® (EVRF®) from F Care Systems (Belgian) for the treatment of primary great and short saphenous vein reflux.

DETAILED DESCRIPTION:
The investigators wish to evaluate its safety, efficacy, and performance. Although it has been shown to be safe and efficacious in its initial trials, these studies have been limited to generally a caucasian-based population, where the vein size, anatomy and distribution of venous incompetence can be different from their asian counterparts. The study will evaluate the technical, anatomical and clinical performance of EVRF® performed on multiple truncal varicose veins, and without mandatory postoperative compression stockings of the GSV, SSV or AASV. The two primary endpoints for this evaluation are technical success at the time of the procedure, and anatomical success, reported as complete closure at 2-weeks, 3 months, 6 months and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age >21 years, able to understand the requirements of the study and provide informed consent.
2. C2 - C5 varicose veins / CVI
3. Symptomatic primaryGSV, SSV or AASV incompetence, with reflux >0.5 seconds on colour duplex, including one or more of the following symptoms: aching, throbbing, heaviness, fatigue, pruritus, night cramps, restlessness, generalized pain or discomfort, swelling.
4. Patients who has GSV, SSV or AASV diameters of 3mm to 12mm in the standing position.

Exclusion Criteria:

1. Current DVT or history of DVT
2. Recurrent varicose veins
3. Pregnant patients
4. Arterial disease (ABPI<0.8)
5. Sepsis
6. Patients who are unwilling to participate
7. Inability or unwillingness to complete questionnaires
8. Adverse reaction to sclerosant or cyanoacrylate
9. GSV, SSV or AASV severely tortuous
10. Life expectancy < 1 year
11. Active treatment for malignancy other than non-melanoma skin cancer
12. Current, regular use of systemic anticoagulation (e.g. warfarin, heparin)
13. Daily use of narcotic analgesia or NSAIDS to control pain associated with venous disease

Ages: 21 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who will be undergoing Endovenous Radio Frequency® (EVRF®) as a treatment for their varicose veins / chronic venous insufficiency
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Technical Success at time of procedure | Immediately post-procedure
  Occlusion of treated vein post-procedure
Anatomical Success | 2 weeks to 12 months post-procedure
  Anatomical success defined as occlusion of treated vessel, as determined by duplex ultrasound.

SECONDARY OUTCOMES:
Quality of Life Score using the EQ-5D questionnaire | 2 weeks, 3 months, 6 months, 12 months post-procedure
  EQ5D is used to assess quality of life based on Mobility, Self-Care, Usual Activities, Pain/Discomfort and Anxiety, rated at 5 levels: no problems, slight problems, moderate problems, severe problems, unable to perform activity. Inputs from this questionnaire is used to observe for changes in quality of life overtime.
Quality of Life Score using the Chronic Venous Insufficiency Questionnaire (CIVIQ) | 2 weeks, 3 months, 6 months, 12 months post-procedure
  CIVIQ is a questionnaire based on three dimensions - pain, physical and psychological, based on a scale from 1 to 5 (no trouble, slight, moderate, considerable, severe). Based on inputs, Global Index Score (GIS) will be tabulated, ranging for 0 to 100 - the higher the value, the poorer the quality of life.
Quality of Life score using the Aberdeen Varicose Vein Questionnaire (AVVQ) | 2 weeks, 3 months, 6 months, 12 months post-procedure
  To measure health status of varicose veins patients based on symptoms and impact on daily activities. A total score ranging from 0 to 100 will be tabulated, with 100 being worst quality of life
Clinical Change using Venous Clinical Severity Score (VCSS) | 2 weeks, 3 months, 6 months, 12 months post-procedure
  VCSS evaluates the severity of hallmarks of venous disease - 0 (none), 1 (mild), 2 (moderate), 3 (severe).
Pain Score | First 10 days post-operation
  Using a numerical rating scale, which ranges from 0 (no pain) to 10 (severe pain)
Time taken to return to work and normal activities | 10 days post-operation
Occlusion rates | 2 weeks, 3 months, 6 months, 12 months post-procedure
  Duplex ultrasound performed at specific timepoints to ensure that treated vein is occluded
Patient satisfaction with treatment: survey | 2 weeks, 3 months, 6 months, 12 months post-procedure
  A short survey to assess patient satisfaction and if there are any observed improvement in terms of appearance and symptoms post-procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Tjun Yip Tang, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapre General Hospital, Singapore, Singaopore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gloviczki P, Comerota AJ, Dalsing MC, Eklof BG, Gillespie DL, Gloviczki ML, Lohr JM, McLafferty RB, Meissner MH, Murad MH, Padberg FT, Pappas PJ, Passman MA, Raffetto JD, Vasquez MA, Wakefield TW; Society for Vascular Surgery; American Venous Forum. The care of patients with varicose veins and associated chronic venous diseases: clinical practice guidelines of the Society for Vascular Surgery and the American Venous Forum. J Vasc Surg. 2011 May;53(5 Suppl):2S-48S. doi: 10.1016/j.jvs.2011.01.079. PMID 21536172
- [Background] Beebe-Dimmer JL, Pfeifer JR, Engle JS, Schottenfeld D. The epidemiology of chronic venous insufficiency and varicose veins. Ann Epidemiol. 2005 Mar;15(3):175-84. doi: 10.1016/j.annepidem.2004.05.015. PMID 15723761
- [Background] van den Bos R, Arends L, Kockaert M, Neumann M, Nijsten T. Endovenous therapies of lower extremity varicosities: a meta-analysis. J Vasc Surg. 2009 Jan;49(1):230-9. doi: 10.1016/j.jvs.2008.06.030. Epub 2008 Aug 9. PMID 18692348
- [Background] Geza M, Gloviczki P. Venous Embryology and Anatomy. In: Bergan JJ, editor. The Vein Book: Elsivier Academic Press; 2007.
- [Background] van Eekeren RR, Boersma D, de Vries JP, Zeebregts CJ, Reijnen MM. Update of endovenous treatment modalities for insufficient saphenous veins--a review of literature. Semin Vasc Surg. 2014 Jun;27(2):118-36. doi: 10.1053/j.semvascsurg.2015.02.002. Epub 2015 Feb 18. PMID 25868763
- [Background] Guex JJ. Endovenous chemical (and physical) treatments for varices: what's new? Phlebology. 2014 May;29(1 suppl):45-48. doi: 10.1177/0268355514526331. Epub 2014 May 19. PMID 24843085
- [Background] Davies HO, Popplewell M, Darvall K, Bate G, Bradbury AW. A review of randomised controlled trials comparing ultrasound-guided foam sclerotherapy with endothermal ablation for the treatment of great saphenous varicose veins. Phlebology. 2016 May;31(4):234-40. doi: 10.1177/0268355515595194. Epub 2015 Jul 9. PMID 26163507